CLINICAL TRIAL: NCT00373516
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Study of the Safety and Efficacy of Two Dosing Regimens of QRX-101 (Becocalcidiol) Ointment in the Treatment of Plaque-Type Psoriasis
Brief Title: Safety and Efficacy Study of Two Dose Regimens of Becocalcidiol in the Treatment of Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QuatRx Pharmaceuticals Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QRX-101-CLIN-003
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Psoriasis
Keywords: psoriasis; topical therapy
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: Vehicle (Placebo) applied BID
Drug: QRX-101 75 mcg/g ointment applied QD
Drug: QRX-101 75 mcg/g ointment applied BID

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two dosing regimens of QRX-101 ointment (75 mcg/g QD and 75mcg/g BID) in the treatment of plaque-type psoriasis when applied topically twice daily for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable plaque-type psoriasis affecting 2% to 10% of the subject's body surface area
* Psoriasis of a severity that is appropriate for treatment with topical therapy; PGA of at least 3 (moderate) at baseline; PSS of at least 7, and with no individual symptom score (erythema, induration, or scaling) less than 2
* Subject must sign the IRB approved informed consent and agree to follow dosing instructions and complete required clinic visits.

Exclusion Criteria:

* Pregnant or nursing females
* Systemic corticosteroids, methotrexate, cyclosporine, systemic retinoids, prolonged sun exposure or ultraviolet light therapy within 4 weeks of dosing
* Topical corticosteroids, retinoids, calcipotriene, coal tar, anthralin, or any other treatment indicated for psoriasis within 2 weeks of dosing
* Untreated bacterial, tubercular, fungal or any viral lesion of the skin
* Biologic agents/monoclonal antibodies in the last 6 months
* Currently using lithium or plaquenil
* Currently using a beta-blocking medication or thiazide diuretic and the dose has not been stabilized for at least 6 months
* History of hypercalcemia or evidence of vitamin D toxicity
* Current or history of melanoma skin cancer in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-09; Study Completion 2005-03

PRIMARY OUTCOMES:
Dichotomized Physician's Static Global Assessment of Overall Lesion Severity (PGA)at Week 8
Percent Change from Baseline in Psoriasis Symptom Severity (PSS)Scale at Week 8

SECONDARY OUTCOMES:
Dichotomized PGA at weeks 2 and 4
Ordinal PGA at weeks 2, 4, and 8
Percent change from baseline PSS at weeks 2 and 4
Ordinal PSS at weeks 2, 4, and 8
Individual symptom scores (erythema, induration, and scaling) at weeks 2, 4, and 8
Body surface area (BSA) involvement at weeks 2, 4, and 8

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Clinical Research Site, Hot Springs, Arkansas
  - Clinical Research Site, Santa Rosa, California
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, Lexington, Kentucky
  - Clinical Research Site, Louisville, Kentucky
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Edina, Minnesota
  - Clinical Research Site, Winston-Salem, North Carolina
  - Clinical Research Site, Temple, Pennsylvania
  - Clinical Research Site, Anderson, South Carolina
  - Clinical Research Site, Simpsonville, South Carolina
  - Clinical Research Site, San Antonio, Texas

REFERENCES:
- [Background] Barker JN, Ashton RE, Marks R, Harris RI, Berth-Jones J. Topical maxacalcitol for the treatment of psoriasis vulgaris: a placebo-controlled, double-blind, dose-finding study with active comparator. Br J Dermatol. 1999 Aug;141(2):274-8. doi: 10.1046/j.1365-2133.1999.02975.x. PMID 10468799
- [Background] Bourke JF, Berth-Jones J, Iqbal SJ, Hutchinson PE. High-dose topical calcipotriol in the treatment of extensive psoriasis vulgaris. Br J Dermatol. 1993 Jul;129(1):74-6. doi: 10.1111/j.1365-2133.1993.tb03315.x. PMID 8369213
- [Background] Bourke JF, Berth-Jones J, Mumford R, Iqbal SJ, Hutchinson PE. High dose topical calcipotriol consistently reduces serum parathyroid hormone levels. Clin Endocrinol (Oxf). 1994 Sep;41(3):295-7. doi: 10.1111/j.1365-2265.1994.tb02548.x. PMID 7955435
- [Background] Bourke JF, Iqbal SJ, Hutchinson PE. Vitamin D analogues in psoriasis: effects on systemic calcium homeostasis. Br J Dermatol. 1996 Sep;135(3):347-54. PMID 8949424
- [Background] Frappaz A, Thivolet J. (1993). Calcipotriol in combination with PUVA: A randomized double-blind placebo study in severe psoriasis. European Journal of Dermatology. 3:351-354.
- [Background] Javitz HS, Ward MM, Farber E, Nail L, Vallow SG. The direct cost of care for psoriasis and psoriatic arthritis in the United States. J Am Acad Dermatol. 2002 Jun;46(6):850-60. doi: 10.1067/mjd.2002.119669. PMID 12063481
- [Background] Krueger G, Koo J, Lebwohl M, Menter A, Stern RS, Rolstad T. The impact of psoriasis on quality of life: results of a 1998 National Psoriasis Foundation patient-membership survey. Arch Dermatol. 2001 Mar;137(3):280-4. PMID 11255325
- [Background] Lamba S, Lebwohl M. Combination therapy with vitamin D analogues. Br J Dermatol. 2001 Apr;144 Suppl 58:27-32. doi: 10.1046/j.1365-2133.2001.144s58027.x. PMID 11501510
- [Background] Lebwohl M, Ali S. Treatment of psoriasis. Part 1. Topical therapy and phototherapy. J Am Acad Dermatol. 2001 Oct;45(4):487-98; quiz 499-502. doi: 10.1067/mjd.2001.117046. PMID 11568737
- [Background] Salmhofer W, Maier H, Soyer HP, Honigsmann H, Hodl S. Double-blind, placebo-controlled, randomized, right-left study comparing calcipotriol monotherapy with a combined treatment of calcipotriol and diflucortolone valerate in chronic plaque psoriasis. Acta Derm Venereol Suppl (Stockh). 2000;(211):5-8. doi: 10.1080/00015550050500022. PMID 11234559
- [Derived] Helfrich YR, Kang S, Hamilton TA, Voorhees JJ. Topical becocalcidiol for the treatment of psoriasis vulgaris: a randomized, placebo-controlled, double-blind, multicentre study. Br J Dermatol. 2007 Aug;157(2):369-74. doi: 10.1111/j.1365-2133.2007.08037.x. Epub 2007 Jun 26. PMID 17596167